CLINICAL TRIAL: NCT00557232
Title: The RAVE (Rubeosis Anit-VEgf) Trial, Utilizes Monthly Intravitreal Bevazizumab (Avastin) Injections for 12 Months to See if Total VEGF Blockade Will Prevent Neovascular Glaucoma and Eliminate the Need for Panretinal Photocoagulation in Patients With Ischemic Central Retinal Vein Occlusion
Brief Title: Intraocular Bevacizumab (Avastin) for Rubeosis Iridis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Principal Investigator, Joao Nassaralla, MD, Instituto de Olhos de Goiania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JN-01-2007-ARVO
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Glaucoma; Rubeosis Iridis
Keywords: bevacizumab; rubeosis iridis; glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bevacizumab — 1.25mg/month

SUMMARY:
Bevacizumab (Avastin®, Roche, Rio de Janeiro, Brazil) is an anti-VEGF recombinant humanized monoclonal IgG1 antibody used to treat colorectal cancers. Bevacizumab may have a role in treating ocular disorders involving fibrovascular proliferation. To determine whether intraocular bevacizumab decreases rubeosis iridis in patients with neovascular glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Ischemic CRVO within 3 months of enrollment as per the following inclusion criteria
* Three of the following clinical tests must be present to demonstrate ischemic CRVO:

  * VA 20/200 or worse
  * RAPD 0.9 LU or worse
  * Loss of 1-2e isopter on Goldmann Visual field (Kwon et al. 2001)
  * ERG demonstrating b wave amplitude less than 60% of A wave

Exclusion Criteria:

* Angle neovascularization greater than 3 clock hours with IOP over 30 (Neovascular glaucoma)
* Any previous retinal laser photocoagulation to the study eye
* Any previous intravitreal injection in study eye (triamcinolone or other)
* Any previous vitrectomy in study eye (posterior or anterior associated with vitreous loss in cataract surgery)
* Intracapsular cataract extraction (posterior capsule needs to be present)
* Previous history of retinal detachment in study eye
* Any previous radiation treatments to head/ neck
* Inability to assess iris neovascularization (corneal opacity precluding gonioscopy)
* Significant cardiovascular disease or cancer that would prevent follow-up visits or completion of the 12 month study
* Significant diabetic retinopathy in the fellow eye (diabetic macular edema, proliferative diabetic retinopathy, or high-risk non-proliferative diabetic retinopathy)
* Pregnancy (positive pregnancy test)
* Prior enrollment in any study for vein occlusion in the study eye
* Participation in another simultaneous medical investigator or trial
* Ocular disorders in the study eye that may confound interpretation of study results, including retinal detachment, macular hole, or choroidal neovascularization of any cause (e.g., DME AMD, ocular histoplasmosis, or pathologic myopia)
* Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the study period
* Aphakia or absence of the posterior capsule in the study eye
* Previous violation of the posterior capsule is also excluded unless it occurred as a result of YAG laser posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation.
* History of idiopathic or autoimmune uveitis in either eye
* Structural damage to the center of the macula in the study eye preexisting to CRVO likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s)
* Vitreomacular traction or epiretinal membrane in the study eye evident biomicroscopically or by OCT
* Ocular inflammation (including trace or above) in the study eye
* Uncontrolled glaucoma (defined as intraocular pressure ≥30 mm Hg despite treatment with anti- medications) or previous filtration surgery in the study eye
* Systemic Conditions
* Uncontrolled Blood pressure exceeding diastolic pressure of 100 mm Hg (sitting) during the screening period
* Uncontrolled diabetes mellitus
* Renal failure requiring dialysis or renal transplant
* Premenopausal women not using adequate contraception
* Previous participation in other studies of investigational drugs (excluding vitamins and minerals) within 3 months preceding Day 0
* History of other disease, metabolic dysfunction, physical examination finding, or other findings giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug, might affect interpretation of the results of the study, or render the subject at high risk from treatment complications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-11; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Intraocular Bevacizumab (Avastin) for Rubeosis Iridis | Compare results
  RI was investigated prospectively by iris biomicroscopy. An expanded informed consent with an off-label use waiver and explanation letter was reviewed with all patients

CONTACTS AND LOCATIONS:
Overall Officials: Joao J Nassaralla, Jr., Principal Investigator — Instituto de Olhos de Goiânia